CLINICAL TRIAL: NCT06820827
Title: Effect of High Power Pain Threshold Ultrasound on Postnatal Sacroiliac Joint Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Hassan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005376
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Sacroiliac Joint Dysfunction
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release group (Active Comparator): The participants will receive myofascial release three times/week for eight weeks.
  Interventions: Other: Myofascial release
- Myofascial release and high-power pain threshold ultrasound group (Experimental): The participants will receive myofascial release in addition to a high-power pain threshold ultrasound on the sacroiliac joint for 20 minutes three times a week for eight weeks.
  Interventions: Other: Myofascial release; Device: High-power pain threshold ultrasound

INTERVENTIONS:
Other: Myofascial release — The participants will receive myofascial release (MFR) on erector spinae, quadratus lumborum, piriformis and gluteus medius. The duration of MFR for each muscle will be 90 to 120 seconds, three times/week for eight weeks.
Device: High-power pain threshold ultrasound — The participants will receive high-power pain threshold ultrasound on sacroiliac joint, 20 minutes, three times/week for eight weeks.
  Arms: Myofascial release and high-power pain threshold ultrasound group

SUMMARY:
This study will be conducted to investigate the effect of high-power pain threshold ultrasound on postnatal sacroiliac joint pain.

DETAILED DESCRIPTION:
Sacroiliac joint pain (SIJ) in the pregnant and postpartum females is susceptible to dysfunction due to multiple biomechanical changes that happen over the course of gestation. This includes an increased angle of lordosis, weight gain, and structural trauma due to the physiologic process of childbirth, biomechanical changes, along with hormonal fluctuations through each trimester, particularly with increased levels of estrogen and relaxin, have been found to decrease the stability of the joint leading to sustained postpartum back pain that may necessitate surgical intervention if conservative treatment fails.

PGP can result in significant physical disability and has important psychosocial implications, including extended leave from work during pregnancy and postnatal, poorer quality of life (as a result of being unable to carry out normal roles, affecting their ability to care for their children and the new baby) and predisposition to chronic pain.

There are side effects to using medical treatment for PGP, such as bruising, bleeding, stomach upset (including bleeding in the stomach), peptic (stomach) ulcers, blurred vision, constipation, dry mouth, fatigue, headaches, insomnia, mood changes, nausea, urination problems, and weight gain. So, using other treatment methods, such as ultrasound therapy to treat PGP is beneficial.

Ultrasound therapy is a non-invasive treatment in which sound waves penetrate soft tissues, increasing blood flow; this can help relieve pain, improve circulation, and promote tissue healing. As such, ultrasound therapy is often used to treat injuries, muscle spasms, and chronic issues like neck or back pain.

No previous study has investigated the effect of high-power pain ultrasound on sacroiliac pain in postpartum women. So, this study aims to investigate the effect of high-power ultrasound on postnatal sacroiliac joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women diagnosed with sacroiliac joint pain and referred by an orthopedist.
* Their ages will range from 20 to 30 years old.
* Their body mass index (BMI) will range from 25 to 29.9 kg/m2.
* All of them should have symptoms for at least two weeks postnatal

Exclusion Criteria:

* Kidney diseases like stones or renal failure
* History of ischemic heart diseases or Myocardial infarction
* Severe vitamin D3 deficiency
* Severe liver diseases or hepatitis
* Psychological distress

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  A numerical rating scale will be used to evaluate pain intensity for all participants before and after the end of the treatment program. It will be given to each participant to rate her intensity of pain. 0 indicates no Pain, 1-3 indicates mild pain (nagging, annoying, interfering little with activity of daily living (ADLs), 4-6 indicates moderate pain (interferes significantly with ADLs), and 7-10 indicates severe pain (disabling; unable to perform ADLs).
Pressure pain threshold (PPT) | 8 weeks
  A pressure algometry (Force Dial model FDK 20 Push Pull Force Gage, Wagner Instruments, Greenwich CT, USA) will be used to assess pain sensitivity by measuring pressure pain thresholds (PPT) at five selected points in the sacroiliac joint region of the affected side. The first examined point will be 1 cm medial and inferior to the posterior superior iliac spine, while the other four examined points will be 2 cm lateral, medial, superior, and inferior to the first point. Each point was measured three times with a ten-second interval between them; the mean of them will be then calculated for each point to be utilized for statistical analysis.

SECONDARY OUTCOMES:
Function disability | 8 weeks
  Pelvic Pain Impact Questionnaire (PPIQ) will be used to assess function disability. It consists of 8 questions that get scored 0-4, for a total of 32. 0 indicates no at all and 4 indicates great deal.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Ali, PHD, Study Director — Cairo University; Doaa Osman, Professor, Study Chair — Cairo University
Locations (1):
- Ahmed Mohamed Mohamed, Cairo, Egypt